CLINICAL TRIAL: NCT01990963
Title: Brain Densitometric Assessment With Axial Computerized Tomography After Severe Brain Trauma.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Paolo Severgnini, Prof., Università degli Studi dell'Insubria
Other Study IDs: 346
Record Dates: First submitted 2013-11-07; First posted 2013-11-25 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Severe Brain Trauma
Keywords: Brain trauma;; MALUNA;; densitometric data; CT
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Processing the Digital Imaging and COmmunications in Medicine (DICOM) of tomographic using Mannheim Lung Analyzing software (MALUNA®) , to obtain volumetrical and densitometric data of brain tissue after patients with severe brain trauma

DETAILED DESCRIPTION:
Quantitative analysis of brain and structures in it, in terms of volume, weight and density, in patients with severe brain trauma, using MALUNA dedicated software to process DICOM images.

1. st endpoint: compare these data with those obtained by CT scans analysis of patients that recur to this kind of diagnostic investigation for non-traumatic events and with negative diagnostic related to cerebral pathological implication.
2. nd endpoint: relate data obtained with clinical evaluation of the patient (cerebral physiology and outcome)
3. rd endpoint: evaluate differences in terms of volume, weight and density of brain and its structures, between patients with diffuse cerebral injury and those with localized lesions.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, any ethnic group
* Patient with severe brain trauma (GCS < 8)
* Need of mechanical ventilation
* Clinical need of urgent CT study of brain.
* Need of clinical control of CT study of brain within first 72 hours from event
* Informed consent obtained from solicitor, due to the fact that patient is

Exclusion Criteria:

* Age minor than 18 yrs old at hospitalization day
* Cardiac arrest pre-hospital or in-hospital and post-anoxic coma
* Non traumatic coma
* Exaggerated ingestion of depressors of central nervous system
* Documented abuse of narcotic drugs;
* Documented abuse of alcohol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female, any ethnic group with severe brain trauma
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2010-01; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
The evaluation of volumetrical and densitometric data of brain tissue of patients with severe brain trauma | Participants will be followed for 8 days

SECONDARY OUTCOMES:
The evaluation of consciousness. | Participants will be followed for 8 days
  During the observation are evaluated:
  • Glasgow Coma Scale (GCS).
The evaluation of clinical conditions. | Participants will be followed for 8 days
  During the observation are evaluated multiparametric arterial and venous gas analysis :
  partial pressure of oxygen in arterial blood(PaO2); partial pressure of carbon dioxide in the arterial blood (PaCO2); cerebral venous oxygen saturation (SjO2); arterial oxygen saturation (SaO2); measure of the acidity or basicity of an aqueous solution (pH); base excess (B.E.); bicarbonate ion (HCO3-); sodium ion (Na+); potassium ion (K+); glycemia; blood concentration of hemoglobin(Hb); hematocrit (Ht).
The evaluation of brain pressures | Participants will be followed for 8 days
  During the observation are evaluating:
  • Intracranial Cerebral Pressure (ICP) if monitored and perfusional cerebral pressure(PCP);
The evaluation of cardiac monitoring. | Participants will be followed for 8 days
  During the observation are evaluating:
  • Mean arterial pressure (MAP), cardiac frequency (FC), body temperature, water balance, diuresis;

CONTACTS AND LOCATIONS:
Overall Officials: Paolo MD Severgnini, Prof., Principal Investigator — Università degli Studi dell'Insubria, Varese, Italia
Locations (1):
- Azienda ospedaliera ospedale Circolo e Fondazione Macchi, Varese, Italy